CLINICAL TRIAL: NCT06992804
Title: The Efficacy and Safety of Near-Infrared Light Therapy Combined With Lecanemab for Mild Alzheimer's Disease
Brief Title: Near-Infrared Light Therapy Combined With Lecanemab for Mild Alzheimer's Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024346
Record Dates: First submitted 2025-03-18; First posted 2025-05-28 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — lecanemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Core phase: Near infrared light therapy with lecanemab (Experimental)
  Interventions: Other: NirsCure with Lecanemab
- Core phase: Sham irradiation with lecanemab (Placebo Comparator)
  Interventions: Other: sham NirsCure with Lecanemab
- Extension phase: Near infrared light therapy with lecanemab (Experimental): This arm includes participants who finish the core phase and are willing to take part in the extension phase.
  Interventions: Other: NirsCure with Lecanemab

INTERVENTIONS:
Other: NirsCure with Lecanemab — Near-infrared light therapy (one session per day, 30 minutes per session, 6 sessions per week) combined with lecanemab (10mg/kg).
  Arms: Core phase: Near infrared light therapy with lecanemab
Other: sham NirsCure with Lecanemab — Sham near-infrared light therapy (where only the equipment appearance is consistent with the true near infrared light device, one session per day, 30 minutes per session, 6 sessions per week) in combined with lecanemab (10mg/kg).
  Arms: Core phase: Sham irradiation with lecanemab
Other: NirsCure with Lecanemab — Near-infrared light therapy (one session per day, 30 minutes per session, 6 sessions per week) combined with lecanemab (10mg/kg).
  Arms: Extension phase: Near infrared light therapy with lecanemab

SUMMARY:
The goal of this study is to explore the efficacy and safety of near-infrared light combined with lecanemab in patients with mild Alzheimer's disease (AD).

This study will employ a randomized, double-blind, sham-controlled method with an open-label extension phase. This trial contains the core phase and an extension phase. During the core phase, eligible subjects were selected and randomized (experimental group: control group = 1:1). The subjects who entered the experimental group received treatment with a near-infrared light therapy device combined with lecanemab for 16 weeks. The subjects who entered the control group received treatment with a near-infrared light therapy device simulator (sham stimulation) combined with lecanemab for 16 weeks. After completing the core phase, patients from both groups of the core phase are eligible to enter the extension phase. In the extension phase, all the participants were treated with a near-infrared light therapy device combined with lecanemab up to week 48.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 50 and 90 years old, gender unrestricted;
2. Meet the core clinical diagnostic criteria for probable Alzheimer's disease as defined by the National Institute on Aging and the Alzheimer's Association (2011 NIA-AA);
3. Amyloid positivity confirmed by Amyloid PET;
4. Clinical Dementia Rating - Global Score (CDR-GS) rating = 1;
5. Mini-Mental State Examination (MMSE) score ≥ 15;
6. Participants must have an educational level of primary school or above and be capable of completing the cognitive assessments and other tests as specified in the protocol;
7. If taking cognition-enhancing medications, the dosage must have been stable for at least 12 weeks prior to enrollment (psychotropic drug dosage stable for at least 4 weeks);
8. The participant or their guardian voluntarily agrees to participate and signs the informed consent form.
9. For caregivers, the following requirements must be met: They need to be stable and have the ability to read. A minimum of 1 hour of daily interaction with the participant is necessary. Throughout the study, they are expected to assist in completing the informant sections of the scale assessments. Additionally, they should be willing to help the participant use the near-infrared light therapy device. Finally, they must understand and agree to the study procedures.

Exclusion Criteria:

1. Cognitive impairment or dementia due to any cause other than Alzheimer's disease, or severe psychiatric disorders (schizophrenia, bipolar disorder, severe depression, etc.);
2. APOE genotype of ε4/ε4;
3. More than 5 cerebral microbleeds in the cerebral cortex as indicated by MRI within the last three months;
4. Currently taking anticoagulant medications;
5. History of epilepsy or hemorrhagic stroke within the past 12 months;
6. Allergy to sunlight or visible light, or high sensitivity of the skin on the head and neck;
7. Severe head trauma or presence of implanted devices (bone screws, bone plates, surgical removals, etc.);
8. Malignant tumors;
9. Any unstable and uncontrolled medical conditions (such as severe cardiac, respiratory, gastrointestinal, renal diseases), or conditions that the investigator deems may affect the safety of the patient or interfere with trial assessments;
10. Contraindications to PET or MRI, including claustrophobia, cardiac pacemaker/defibrillator, ferromagnetic metal implants, etc.;
11. Currently receiving anti-amyloid treatment for Alzheimer's disease with severe adverse reactions such as cerebral hemorrhage or cerebral edema;
12. Alcohol or drug addiction;
13. Pregnant, breastfeeding, or planning to become pregnant;
14. Participation in another clinical study within one month prior to this trial;
15. Other situations deemed by the investigator as unsuitable for participation in the clinical study.
16. For caregivers, the following exclusion criterion applies: They must not have severe neurological or psychiatric disorders.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in the Alzheimer's Disease Assessment Scale-Cognitive (ADAS-cog). | 16 weeks.
  The Alzheimer's Disease Assessment Scale - Cognitive Section (ADAS-Cog-14) is a comprehensive tool used to evaluate cognitive function in individuals. The unabbreviated scale title is the Alzheimer's Disease Assessment Scale - Cognitive Section. The minimum score on this scale is 0, while the maximum score is 144. Importantly, higher scores on the ADAS-Cog-14 indicate worse cognitive function. This scale assesses various cognitive domains, and an increasing score reflects more severe cognitive impairment.

SECONDARY OUTCOMES:
The change from baseline in the Alzheimer's Disease Assessment Scale-Cognitive (ADAS-cog). | 32 weeks, 48 weeks.
  The Alzheimer's Disease Assessment Scale - Cognitive Section (ADAS-Cog-14) is a comprehensive tool used to evaluate cognitive function in individuals. The unabbreviated scale title is the Alzheimer's Disease Assessment Scale - Cognitive Section. The minimum score on this scale is 0, while the maximum score is 144. Importantly, higher scores on the ADAS-Cog-14 indicate worse cognitive function. This scale assesses various cognitive domains, and an increasing score reflects more severe cognitive impairment.
The change from baseline in the Mini-Mental State Examination (MMSE). | 16 weeks, 32 weeks, 48 weeks.
  The Mini-Mental State Examination (MMSE) is a widely used tool for assessing cognitive function. The unabbreviated scale title is the Mini-Mental State Examination. The minimum score on this scale is 0, while the maximum score is 30. Higher scores on the MMSE indicate better cognitive function. This scale evaluates various cognitive domains such as orientation, attention, calculation, recall, and language. A higher score reflects better cognitive performance.
The change from baseline in the Clinical Dementia Rating - Sum of Boxes (CDR-SB). | 16 weeks, 32 weeks, 48 weeks.
  The Clinical Dementia Rating - Sum of Boxes (CDR-SB) is a comprehensive assessment tool used to evaluate the severity of dementia. The unabbreviated scale title is the Clinical Dementia Rating - Sum of Boxes. The minimum score on this scale is 0, while the maximum score is 18. Higher scores on the CDR-SB indicate worse cognitive and functional impairment. This scale assesses various domains including memory, orientation, judgment and problem-solving, community affairs, home and hobbies, and personal care. An increasing score reflects more severe dementia.
The change from baseline in the Alzheimer's Disease Cooperative Study - Activities of Daily Living Scale (ADCS-ADL). | 16 weeks, 32 weeks, 48 weeks.
  The Alzheimer's Disease Cooperative Study - Activities of Daily Living Scale (ADCS-ADL) is a tool designed to assess the functional abilities of individuals in their daily activities. The unabbreviated scale title is the Alzheimer's Disease Cooperative Study - Activities of Daily Living Scale. The minimum score on this scale is 0, while the maximum score is 78. Higher scores on the ADCS-ADL indicate better functional ability in daily living activities. This scale evaluates various aspects of daily living, such as personal care, household chores, and financial management. A higher score reflects better performance in activities of daily living.
The change from baseline in the Neuropsychiatric Inventory (NPI). | 16 weeks, 32 weeks, 48 weeks.
  The Neuropsychiatric Inventory (NPI) is a comprehensive assessment tool used to evaluate behavioral and psychiatric symptoms in individuals with cognitive disorders. The unabbreviated scale title is the Neuropsychiatric Inventory. The minimum score on this scale is 0, while the maximum score is 144. Higher scores on the NPI indicate more severe behavioral and psychiatric symptoms. This scale assesses various domains including delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, euphoria/elation, apathy/indifference, disinhibition, irritability/lability, and motor disturbance. An increasing score reflects more significant behavioral and psychiatric disturbances.
The change from baseline in the Hamilton Depression Rating Scale (HAMD). | 16 weeks, 32 weeks, 48 weeks.
  The Hamilton Depression Rating Scale (HAMD) is a widely used tool for assessing the severity of depressive symptoms in individuals. The unabbreviated scale title is the Hamilton Depression Rating Scale. The minimum score on this scale is 0, while the maximum score is 52 (for the 17-item version). Higher scores on the HAMD indicate more severe depressive symptoms. This scale evaluates various aspects of depression, including mood, guilt, suicide, insomnia, agitation, anxiety, somatic symptoms, and weight loss. An increasing score reflects more significant depressive symptomatology.
The change from baseline in the Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC). | 16 weeks, 32 weeks, 48 weeks.
  The Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) is a tool used to assess the overall change in clinical status of individuals with Alzheimer's disease. The unabbreviated scale title is the Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change. The scale ranges from 1 to 7, with 1 indicating "Very much improved" and 7 indicating "Very much worse." A score of 4 represents "No change." Lower scores on the ADCS-CGIC indicate better clinical outcomes, reflecting improvement or stabilization, while higher scores indicate worsening clinical status. This scale provides a global assessment of change based on the clinician's judgment of the patient's overall condition.
The change from baseline levels measured by Positron Emission Tomography (PET). | 16 weeks, 48 weeks.
The change from baseline as measured by Magnetic Resonance Imaging (MRI). | 16 weeks, 32 weeks, 48 weeks.
The change from baseline in blood biomarker measurements. | 16 weeks, 32 weeks, 48 weeks.
  Concentration of Abeta-40, Abeta-42, t-tau, p-tau181, p-tau217, GFAP, NFL
The change from baseline as measured by EEG power across different frequency bands. | 16 weeks, 32 weeks, 48 weeks.
  This outcome measure assesses changes in EEG power across different frequency bands, including Delta (1-4 Hz), Theta (4-8 Hz), Alpha (8-12 Hz), Beta (12-30 Hz), and Gamma (30-100 Hz). EEG recordings will be taken at baseline and at specified time points during the study to evaluate changes in brain activity.
  Power: µV²/Hz
  Higher power in specific frequency bands may indicate increased brain activity, while lower power may suggest decreased activity. The clinical significance of changes in EEG power will be interpreted based on the study objectives and relevant clinical standards.
Safety indicators/adverse events. | 16 weeks, 32 weeks, 48 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Tang, MD, PhD, Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No